CLINICAL TRIAL: NCT03552575
Title: The Effects of Sacubitril/Valsartan Compared to Valsartan on Left Ventricular Remodelling in Asymptomatic Left Ventricular Systolic Dysfunction After Myocardial Infarction: a Randomised, Double-blinded, Active-comparator, Cardiac-MR Based Trial
Brief Title: The Effects of Sacubitril/Valsartan Compared to Valsartan on LV Remodelling in Asymptomatic LV Systolic Dysfunction After MI
Acronym: RECOVER-LV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN16CA007
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
Keywords: sacubritil; valsartan; left ventricular remodelling; asymptomatic left ventricular systolic dysfunction; myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, active-comparator, double-blinded study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/valsartan (Experimental): 24mg/26mg (dose level 1), 49mg/51mg (dose level 2) and 97mg/103mg (dose level 3) twice daily
  Interventions: Drug: sacubitril/valsartan
- Valsartan (Experimental): 40mg (dose level 1), 80mg (dose level 2) and 160mg (dose level 3) twice daily.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril is a prodrug neprilysin inhibitor used in combination with valsartan to reduce the risk of cardiovascular events in patients with chronic heart failure (NYHA Class II-IV) and reduced ejection fraction.
  Arms: Sacubitril/valsartan
Drug: Valsartan — is an angiotensin II receptor antagonist (commonly called an ARB, or angiotensin receptor blocker), that is selective for the type I (AT1) angiotensin receptor.
  Arms: Valsartan

SUMMARY:
Prior to reperfusion therapy, the major therapeutic breakthrough in myocardial infarction was the demonstration that ACE inhibitors or ARBs, given to prevent adverse "remodelling" (progressive dilatation and decline in systolic function) in high risk patients, reduced the likelihood of developing heart failure and the risk of death. The neurohumoral systems which are activated in patients after myocardial infarction (and in heart failure) are not all harmful and some endogenous systems may be protective. The best recognised of these is the natriuretic peptide system.

A- and B-type natriuretic peptides are secreted by the heart when it is stressed and these peptides promote vasodilation (reducing left ventricular wall stress), stimulate renal sodium and water excretion (i.e. antagonising the retention of salt and water characterising heart failure) and inhibit pathological growth i.e. hypertrophy and fibrosis (key components of the adverse left ventricular remodelling that occurs after infarction and in heart failure).The augmentation of plasma levels of endogenous natriuretic peptides can be achieved through inhibition of neutral endopeptidase, also known as neprilysin (NEP), which is responsible for the breakdown of natriuretic peptides. Recently, the addition of neprilysin inhibition to blockade of the RAAS (using sacubitril/valsartan), compared with RAAS blockade alone, reduced the risk of heart failure hospitalisation and death in patients with HF-REF. These exciting findings may lead to a new approach to the treatment of heart failure, with an angiotensin receptor neprilysin inhibitor (ARNI) replacing an ACE inhibitor as one of the fundamental treatments for this condition. We believe that the same approach may be beneficial in highrisk survivors of myocardial infarction. Recently, sacubitril/valsartan was shown to ameliorate adverse left ventricular remodelling in an experimental model of acute myocardial infarction. The objective of the present proposal is to gather "proof-ofconcept", mechanistic, evidence in humans to support adoption of this new approach in patients at high risk after myocardial infarction as a result of residual left ventricular systolic dysfunction.

DETAILED DESCRIPTION:
The objective of the present proposal is to obtain information, which is currently not available, on the cardiac effects of sacubitril/valsartan in patients with LVSD, better characterise the neurohumoral actions of sacubitril/valsartan and gather "proof-ofconcept", mechanistic, evidence in humans to support adoption of this new treatment in patients at high risk after myocardial infarction as a result of residual LVSD.

Surprisingly, there is currently limited evidence about how sacubitril/valsartan works in humans. PARADIGM-HF was a large pragmatic mortality/morbidity trial with no mechanistic sub-studies and this is also true of a ongoing trial (PARADISE-MI) in acute myocardial infarction. Moreover, both trials either used or will use an ACE inhibitor (enalapril and ramipril, respectively), rather than an ARB as the active comparator for sacubitril/valsartan; use of valsartan in our study will allow us to precisely define the effects of neprilysin inhibition. A-type (or atrial) natriuretic peptide (ANP), C-type natriuretic peptide (CNP) and adrenomedullin are substrates for neprilysin and may play a role in the action of sacubitril/valsartan but have not been measured in existing clinical trials (in part because of the instability of these peptides and unfeasibility of measuring them in multi-centre, multi-national trials).

Indeed, ANP and CNP are more specific substrates for neprilysin than BNP. As has been mentioned above, cardiac fibrosis appears to be important in the process of LV remodelling in patients with asymptomatic LVSD and the development of HF-REF and is reflected in circulating biomarkers which may be influenced by sacubitril/valsartan

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction (AMI) at least 3 months prior to recruitment

  * Left ventricular ejection ≤40% as measured by transthoracic echocardiography
  * Ability to provide written, informed consent
  * Age ≥18 years
  * Tolerance of a minimum dose of ACE inhibitor/ARB (ramipril 2.5mg BD or equivalent)
  * Treatment with a beta-blocker unless not tolerated or contraindicated.

Exclusion Criteria:

* Contraindication to CMR (ferrous prosthesis, implantable cardiac device or severe claustrophobia)

  * Clinical and/or radiological heart failure (NYHA≥2)
  * Symptomatic hypotension and/or systolic blood pressure <100mmHg
  * eGFR < 30 mL/min/1.73m2 and/or serum potassium >5.2mmol/L
  * Persistent/permanent atrial fibrillation
  * History of AMI within last 3 months
  * History of hypersensitivity or allergy to ACE-inhibitors/ARB
  * History of angioedema
  * Known hypersensitivity to the active study drug substances, contrast media or any of the excipients
  * Obesity (where body girth exceeds MRI scanner diameter)
  * Pregnancy, planning pregnancy, or breast feeding
  * Inability to give informed consent or comply with study protocol
  * Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x ULN at Visit 1, history of hepatic encephalopathy, history of oesophageal varices, or history of portacaval shunt
  * History of biliary cirrhosis and cholestasis
  * Active treatment with cholestyramine or colestipol resins
  * Active treatment with lithium or direct renin inhibitor
  * Participation in another intervention study involving a drug or device within the past 90 days (co-enrolment in observational studies is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McMurray, MBChB PhD, Principal Investigator — NHS GGC and Glasgow University
Locations (2):
- United Kingdom (2):
  - Glasgow Cardiovascular Research Centre, Glasgow, Scotland
  - Glasgow Clinical Research Facility, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brum WS, Docherty KF, Ashton NJ, Zetterberg H, Hansson O, McMurray JJV, Blennow K. Effect of Neprilysin Inhibition on Alzheimer Disease Plasma Biomarkers: A Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2024 Feb 1;81(2):197-200. doi: 10.1001/jamaneurol.2023.4719. PMID 38109077
- [Derived] Docherty KF, Campbell RT, Brooksbank KJM, Dreisbach JG, Forsyth P, Godeseth RL, Hopkins T, Jackson AM, Lee MMY, McConnachie A, Roditi G, Squire IB, Stanley B, Welsh P, Jhund PS, Petrie MC, McMurray JJV. Effect of Neprilysin Inhibition on Left Ventricular Remodeling in Patients With Asymptomatic Left Ventricular Systolic Dysfunction Late After Myocardial Infarction. Circulation. 2021 Jul 20;144(3):199-209. doi: 10.1161/CIRCULATIONAHA.121.054892. Epub 2021 May 13. PMID 33983794

RESULTS

PARTICIPANT FLOW:
Groups:
- Sacubitril/Valsartan: 24mg/26mg, 49mg/51mg and 97mg/103mg twice daily
  sacubitril/valsartan: Sacubitril is a prodrug neprilysin inhibitor used in combination with valsartan to reduce the risk of cardiovascular events in patients with chronic heart failure (NYHA Class II-IV) and reduced ejection fraction. Used in line with SmPC guidelines. Following randomization the aim should be to up-titrate patients to target study drug dose 97/103mg twice daily after 4 weeks . Slower up-titration was permitted if necessary to ensure patient safety and tolerability. Patients will be allowed to stay at dose level 1 or 2 as maintenance dose however efforts should be made to maintain patients on the target dose level 3 or maximally tolerated dose level for as long a duration as possible during the trial. Adjustments to study drug dose level should be based on safety and tolerability with a focus on a) symptomatic hypotension, b) clinically significant decline in renal function and c) hyperkalaemia.
- Valsartan: 40mg, 80mg and 160mg twice daily.
  Valsartan: is an angiotensin II receptor antagonist (commonly called an ARB, or angiotensin receptor blocker), that is selective for the type I (AT1) angiotensin receptor. Used within SmPC guidelines. Following randomization the aim should be to up-titrate patients to target study drug dose 160mg twice daily after 4 weeks . Slower up-titration was permitted if necessary to ensure patient safety and tolerability. Patients will be allowed to stay at dose level 1 or 2 as maintenance dose however efforts should be made to maintain patients on the target dose level 3 or maximally tolerated dose level for as long a duration as possible during the trial. Adjustments to study drug dose level should be based on safety and tolerability with a focus on a) symptomatic hypotension, b) clinically significant decline in renal function and c) hyperkalaemia.
Period: Overall Study
Arm/Group | Sacubitril/Valsartan | Valsartan
Started | 47 | 46
Completed | 46 | 46
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan | Valsartan | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 31 | 57
  >=65 years | 21 | 15 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.6) | 59.7 (10.1) | 60.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 42 | 43 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 44 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End Systolic Volume Index
Description: Change in indexed left ventricular end-systolic volume (LVESVI) measured by cardiac MR measured in ml/m2
Time Frame: baseline and 12 months
Population: There were 3 patients with incomplete data (1 death and 2 did not tolerate the MRI scan) accounting for the difference in overall number of participants randomised to those analyzed.
Measure: Mean (Standard Deviation); unit: ml/m^2
Groups:
- Sacubitril/Valsartan: 24mg/26mg , 49mg/51mg and 97mg/103mg twice daily
  sacubitril/valsartan: Sacubitril is a prodrug neprilysin inhibitor used in combination with valsartan to reduce the risk of cardiovascular events in patients with chronic heart failure (NYHA Class II-IV) and reduced ejection fraction.
- Valsartan: 40mg , 80mg and 160mg twice daily.
  Valsartan: is an angiotensin II receptor antagonist (commonly called an ARB, or angiotensin receptor blocker), that is selective for the type I (AT1) angiotensin receptor.
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 44
ml/m^2 | -4.0 (6.6) | -2.0 (7.3)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.19, Regression, Linear; Adjusted for randomized treatment, baseline value of the outcome, use of diuretics at baseline and time from randomization to cardiac MRI; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.8 to 1.0]

2. Secondary Outcome: Change in N-terminal Prohormone of B-type Natriuretic Peptide Levels
Description: measured in pg/ml
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 46
pg/mL | -39 [-131 to 12] | -21 [-104 to 23]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.31, Regression, Linear; Adjusted for randomized treatment, baseline value of the outcome, and use of diuretics at baseline; Ratio of adjusted geometric means = 0.85, 95% CI 2-sided [0.63 to 1.16]

3. Secondary Outcome: Change in High Sensitivity Troponin I Levels
Description: measured in ng/L
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 46
ng/L | -1.1 [-2.4 to -0.1] | -0.4 [-2.4 to 0.9]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.41, Regression, Linear; Adjusted for randomized treatment, baseline value of the outcome, and use of diuretics at baseline; Ratio of adjusted geometric means = 0.87, 95% CI 2-sided [0.62 to 1.22]

4. Secondary Outcome: Change in Left Ventricular End-Diastolic Volume Index
Description: Change in indexed left ventricular end-diastolic volume (LVEDVI) measured by cardiac MR measured in ml/m2
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 44
ml/m^2 | -4.4 (8.8) | -1.2 (8.6)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.10, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-6.8 to 0.6]

5. Secondary Outcome: Change in Left Atrial Volume Index
Description: Change in indexed Left Atrial Volume (LAVI) measured by cardiac MR measured in ml/m2
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 43
ml/m^2 | -2.8 (9.0) | -0.8 (11.7)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.29, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-6.6 to 2.0]

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction
Description: Change in left ventricular ejection fraction (LVEF) measured by cardiac MR measured in percentage
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: Ejection fraction %
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 44
Ejection fraction % | 1.1 (3.4) | 1.4 (3.6)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.46, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.0 to 0.9]

7. Secondary Outcome: Change in Left Ventricular Mass Index
Description: Change in indexed left ventricular mass (LVMI) measured by cardiac MR measured in grams/m2
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 44
g/m^2 | -2.4 (4.9) | -1.1 (5.0)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.16, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.5 to 0.6]

8. Secondary Outcome: Change in Patient Well Being as Assessed by Patient Global Assessment Questionnaire
Description: Change in patient well being as assessed by patient global assessment questionnaire which is a patient reported outcome measure that involves a patients own response to questions about their overall health and/or disease activity
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 46 | 46
Participants
  Markedly improved | 8 | 8
  Moderately improved | 9 | 7
  Slightly improved | 5 | 10
  Unchanged | 24 | 21
  Slightly worsened | 0 | 0
  Moderately worsened | 0 | 0
  Markedly worsened | 0 | 0
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; Test type: Superiority; p = 0.56, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year of study follow up whilst taking study drug and an additional 30 days following the final study visit.
Arm/Group | Sacubitril/Valsartan | Valsartan
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 8/47 | 1/46
Other Adverse Events (participants affected / at risk) | 12/47 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacubitril/Valsartan (N=47) | Valsartan (N=46)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacubitril/Valsartan (N=47) | Valsartan (N=46)
Worsening renal function or acute kidney injury (Renal and urinary disorders) | 5 (5) | 4 (4)
Hyperkalaemia (Renal and urinary disorders) | 2 (3) | 1 (1)
Symptomatic hypotension (Cardiac disorders) | 7 (8) | 1 (1)
Symptomatic hypotension with systolic blood pressure <90mmHg (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angioedema (Immune system disorders) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03552575/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT03552575/SAP_001.pdf